CLINICAL TRIAL: NCT01690455
Title: Non-interventional Study to Assess the Efficacy of Mircera for Renal Anemia Correction in Dialysis Patients in Everyday Clinical Practice in Poland.
Brief Title: An Observational Study of Mircera in Renal Anemia Correction In Dialysed Patients During Daily Clinical Practice
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25701
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational, multi-center study will evaluate the efficacy and safety of Mircera (methoxy polyethylene glycol-epoetin beta) in renal anemia correction in dialysed patients in daily clinical practice. Patient will receive Mircera according to local summary of product characteristics. Data will be collected for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Adequate iron status
* Signed informed consent form

Exclusion Criteria:

* Anemia due to non-renal causes
* Where investigator considers the patient unsuitable for inclusing for other reasons (e.g. severe co-morbidities as active bleeding, infections or cancer)
* Pregnant or lactating female patients
* Any contraindications against treatment with Mircera (according to local Summary of Product Characteristics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal anemia and on dialysis therapy
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve a hemoglobin level of >/=10 g/dl | 12 months

SECONDARY OUTCOMES:
Safety: incidence of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- Poland (32):
  - Bartoszyce
  - Bydgoszcz
  - Ciechanów
  - Częstochowa
  - Dębica
  - Gliwice
  - Gmina Świecie
  - Gorzów Wielkopolski
  - Grudziądz
  - Hajnówka
  - Jastrzębie Zdrój
  - Jaworzno
  - Kępno
  - Konin
  - Kościerzyna
  - Lodz
  - Milicz
  - Piła
  - Polanica-Zdrój
  - Radom
  - Rybnik
  - Rzeszów
  - Sandomierz
  - Siedlce
  - Starachowice
  - Suwałki
  - Słupsk
  - Warsaw
  - Wołomin
  - Wroclaw
  - Zgorzelec
  - Łapy